CLINICAL TRIAL: NCT04445779
Title: Q10 Preloading Before Cardiac Surgery for Kidney Failure Reduction
Acronym: PREKARKID-10
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Hospital Center, Split (Other)
Responsible Party: Principal Investigator, Hrvoje Vučemilović, Hrvoje Vučemilović, Principal Investigator, Clinical Hospital Center, Split
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 28878529
Record Dates: First submitted 2020-06-05; First posted 2020-06-24 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Acute Kidney Injury; Acute Kidney Failure
MeSH Terms: conditions — Acute Kidney Injury | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CoQ10 (Experimental): Patients will receive per-orally 10 mg/kg of body weight of coenzyme Q10 in the form of Myokinon (PharmaNord, Denmark) in three divided doses. They will receive therapy for at least 10 days before the surgical procedure.
  Interventions: Dietary Supplement: Coenzyme Q10
- Placebo (Placebo Comparator): Patients will receive per-orally placebo in three divided doses.
  Interventions: Dietary Supplement: Coenzyme Q10

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — Patients will receive per-orally 10 mg/kg of body weight of coenzyme Q10 in form of Myokinon (PharmaNord, Denmark) in three divided doses. They will receive therapy for at least 10 days before surgical procedure.

SUMMARY:
Coenzyme Q10 (CoQ10) is an essential molecule in human body. It acts as an antioxidant, a co-factor for energy conversion in mitochondria and has anti-inflammatory effects capable of improving endothelial function. Our goal is to investigate whether CoQ10 is capable to reduce the incidence of acute kidney injury/failure following cardiac surgery. Cardiac surgery is major risk factor for acute kidney injury/failure (AKI/F).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective cardiac surgery

Exclusion Criteria:

* patients receiving high dose vitamin B supplementation (defined as more that 200% of recommended daily allowances)
* patients under warfarin therapy
* urgent surgery
* end stage kidney disease
* therapy with multiple nephrotoxic drugs
* chronic kidney disease
* obstructive uropathy
* previous cardiac surgery procedure
* alcohol abuse
* malignancy
* allergy to any ingredient of Myoqinon capsule
* patients receiving Myoqinon and fail to demonstrate a significant increase in blood concentration of Q10
* uncontrolled hypertension

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Difference in serum creatinine after cardiac surgery indicating kidney injury. | 7 days
  Increase in serum creatinine as defined by KDIGO stages will be used as indicator of kidney injury.
Difference in urinary low molekular weight alpha 1 microglobulin as an indicator of kidney tubular injury. | 3 days
  Alpha 1 microglobulin is an indicator of kidney tubular damage, measured in urine.
Daily urine output during the 72 hours postoperatively. | 3 days
  Urine output less than 0.5 ml/kg/h during 6 hours indicates increased risk of developing AKI.

SECONDARY OUTCOMES:
Length of stay in intensive care unit | 10 days
  Length of stay in intensive care unit will be compared between an intervention and placebo arm of trial.
Advanced glycation endproducts | 7 days
  Elevated advanced glycation endproducts (AGE) in skin, measured using skin autofluorescence, are reliable predictors of cardiovascular disease and diabetes mellitus. Elevated levels before cardiac surgery should also predict increased risk of intraoperative morbidity, mortality and postoperative complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Center Split, Split, Split-Dalmatia County, Croatia